CLINICAL TRIAL: NCT01675999
Title: PRODIGE 22-ECKINOXE : Randomized Phase II Trial of Neoadjuvant FOLFOX 4 Versus FOLFOX 4 With Cetuximab Versus Immediate Surgery in Locally Advanced Colon Cancer
Brief Title: Trial of Neoadjuvant Chemotherapy in Locally Advanced Colon Cancer
Acronym: ECKINOXE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Federation Francophone de Cancerologie Digestive (Other); UNICANCER (Other); Association de Recherche Experimentale et Clinique en Chirurgie Digestive (Other); Association Européenne de Recherche en Oncologie (Other); Merck Serono S.A., Geneva (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P100131
Record Dates: First submitted 2012-02-02; First posted 2012-08-30 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2012-01

CONDITIONS: Colon Cancer; Locally Advanced Malignant Neoplasm
Keywords: Neoadjuvant chemotherapy; Locally advanced malignant neoplasm; colon cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Perioperative simplified FOLFOX-4 chemotherapy
  - Simplified FOLFOX-4 (IV oxaliplatin given over 120 min at a dose of 85 mg/m2 on day 1 followed by IV leucovorin 400 mg/m2 over 2h, IV bolus 5-FU 400 mg/m2 and IV infusional 5-FU 2400 mg/m2 over 46h) for 4 cycles followed by colectomy (3 to 5 weeks after) followed by simplified FOLFOX-4 (8 cycles).
  Interventions: Other: Perioperative simplified FOLFOX-4 chemotherapy
- 2 (Experimental): Perioperative FOLFOX4+Cetuximab chemotherapy Simplified FOLFOX-4 (IV oxaliplatin given over 120 min at a dose of 85 mg/m2 on day 1 followed by IV leucovorin 400 mg/m2 over 2h, IV bolus 5-FU 400 mg/m2 and IV infusional 5-FU 2400 mg/m2 over 46h)+ Cetuximab (IV 500 mg/m2 every 2 weeks) for 4 cycles followed by colectomy (3 to 5 weeks after), followed by simplified FOLFOX-4 + Cetuximab (8 cycles).
  Interventions: Other: Perioperative FOLFOX4+Cetuximab chemotherapy
- 3 (Other): Surgery followed by FOLFOX4 chemotherapy No preoperative chemotherapy Colectomy (maximum 4 weeks after randomization) followed by simplified FOLFOX-4 (IV oxaliplatin given over 120 min at a dose of 85 mg/m2 on day 1 followed by IV leucovorin 400 mg/m2 over 2h, IV bolus 5-FU 400 mg/m2 and IV infusional 5-FU 2400 mg/m2 over 46h) for 12 cycles.
  Interventions: Other: Surgery followed by FOLFOX4 chemotherapy

INTERVENTIONS:
Other: Perioperative simplified FOLFOX-4 chemotherapy — Preoperative chemotherapy
  Arms: 1
Other: Perioperative FOLFOX4+Cetuximab chemotherapy — Preoperative chemotherapy
  Arms: 2
Other: Surgery followed by FOLFOX4 chemotherapy — Preoperative chemotherapy
  Arms: 3

SUMMARY:
In patients with locally advanced colon cancer (high risk stage II and stage III), curative surgery followed by adjuvant FOLFOX-4 chemotherapy has become the standard of care. However, for 30-40% of these patients, the current curative treatment strategy of surgical excision followed by adjuvant chemotherapy fails either to clear locoregional spread or to eradicate distant micrometastases, leading to disease recurrence. Preoperative chemotherapy is an attractive concept for locally advanced colon cancer and has the potential to impact upon both of these causes of failure. Optimum systemic therapy at the earliest possible opportunity may be more effective at eradicating distant metastases than the same treatment given after the delay and immunological stress of surgery. Added to this, shrinking the primary tumor before surgery may reduce the risk of incomplete surgical excision, and the risk of tumor cell shedding during surgery.

ECKINOXE is a multicenter randomized phase II trial designed to evaluate efficacy (response rate) and feasibility (safety, tolerance) of these two chemotherapy regimens (FOLFOX-4 alone and FOLFOX-4+Cetuximab) in a neoadjuvant strategy in patients with locally advanced colon cancer. Control arm includes patients for whom standard treatment comprises surgery followed by adjuvant FOLFOX-4 chemotherapy. This phase II study will assess the feasibility of a neoadjuvant strategy in these patients and determine which neoadjuvant regimen is the most effective in terms of response rate.

DETAILED DESCRIPTION:
See Synopsis below

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed colon adenocarcinoma (≥ 15 cm from the anal verge)
* Assessment of RAS status of the primary colon cancer on biopsies (WT or mutated)
* Colon cancer classified: poor prognosis T3 (T3 bad) - T4 and/ or N2 by abdominal CT scan.
* Non metastatic colon cancer (lung, liver, peritoneal)
* Non complicated primary tumor (obstruction, perforation, bleeding), patients with cancer treated by stomie de derivation may be included in the study.

DPD deficency

* Absence of synchronous colorectal cancer
* Age ≥ 18 years and < 76 years
* ECOG performance status 0-1
* No prior chemotherapy within the last 5 years
* No prior abdominal or pelvic irradiation within the last 5 years
* Life expectancy of 5 years or more
* No history of colorectal cancer within the last 5 years
* Patients with childbearing potential should use effective contraception during the study and the following 6 months
* White blood cell count of 3 x 109/L or more with neutrophils of1.5 x 109/L or more, platelet count of 100 x 109/L or more, hemoglobin of 9 g/dL (5,6 mmol/l) or more
* Total bilirubin of 1.5 x ULN (upper limit of normal) or less
* ASAT and ALAT of 2.5 x ULN or less
* Alkaline phosphatase of 1.5 x ULN or less
* Serum creatinine of 1.5 x ULN or less
* Signed written informed consent obtained prior to any study specific screening procedures

Exclusion Criteria:

* contra-indication to iodinated contrast medium injection including allergy to iodinated contrast medium and renal insufficiency proscribing iodinated injection
* Age > 70 years
* Rectal cancer located within 15 cm from the anal verge by endoscopy or under the peritoneal reflection at surgery or having received radiation therapy prior to surgery
* Complicated primary colon cancer (obstruction, bleeding, perforation)
* Synchronous colorectal cancer
* Metastatic spread at baseline assessment (lung, liver, peritoneal)
* History or current evidence on physical examination of central nervous system disease or peripheral neuropathy ≥ grade 1 Common Toxicity Criteria for Adverse Events (CTCAE) v.3.0
* Known hypersensitivity reaction to any of the components of study treatments
* Presence of inflammatory bowel disease
* HNPCC syndrome or polyposis
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to study treatment start. Incompletely healed wounds or anticipation of the need for major surgical procedure during the course of the study
* Clinically relevant coronary artery disease or history of myocardial infarction in the last 12 months, or high risk of uncontrolled arrhythmia
* Pregnancy (absence to be confirmed by ß-hCG test) or breast-feeding period
* Previous malignancy in the last 5 years
* Medical, geographical, sociological, psychological or legal conditions that would not permit the patient to complete the study or sign informed consent
* Any significant disease which, in the investigator's opinion, would exclude the patient from the study.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2012-05; Primary Completion 2012-05 (Actual); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Histological tumor response in the primary tumor according to the simplified Tumor Regression Grade (TRG) of Ryan | 2 years
  This primary outcome will be evaluated on the surgical specimens: Immediately after surgery (arm C) or after neoadjuvant chemotherapy (4 cycles) and surgery (arms A and B)

SECONDARY OUTCOMES:
Safety and tolerability and efficacy of the neoadjuvant chemotherapy | 9 years
  * Tolerability of the neoadjuvant therapies. SAFETY ISSUE
  * Postoperative morbidity at 60 days. SAFETY ISSUE
•Disease free survival and regression free survival at 3 years | 3 years
•Overall survival at 6 and 7 years | 6 and 7 years
•Quality of life (EORTC QLQ-C30, QLQ-CR29) | 5 years
•Quality and radicality of the surgical excision | 2 years
•Accuracy of pre-treatment CT scan staging and evaluation of radiological response to chemotherapy | 2 years
•Correlation between radiological and histological response | 2 years
•Evaluation of another histopathological grade | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: mehdi karoui, PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Henri Mondor, Paris, France

REFERENCES:
- [Derived] Karoui M, Gallois C, Piessen G, Legoux JL, Barbier E, De Chaisemartin C, Lecaille C, Bouche O, Ammarguellat H, Brunetti F, Prudhomme M, Regimbeau JM, Glehen O, Lievre A, Portier G, Hartwig J, Goujon G, Romain B, Lepage C, Taieb J; for PRODIGE 22 investigators/Collaborators. Does neoadjuvant FOLFOX chemotherapy improve the prognosis of high-risk Stage II and III colon cancers? Three years' follow-up results of the PRODIGE 22 phase II randomized multicentre trial. Colorectal Dis. 2021 Jun;23(6):1357-1369. doi: 10.1111/codi.15585. Epub 2021 Mar 10. PMID 33580623
- [Derived] Karoui M, Rullier A, Piessen G, Legoux JL, Barbier E, De Chaisemartin C, Lecaille C, Bouche O, Ammarguellat H, Brunetti F, Prudhomme M, Regimbeau JM, Glehen O, Lievre A, Portier G, Hartwig J, Goujon G, Romain B, Lepage C, Taieb J; for PRODIGE 22 investigators/collaborators. Perioperative FOLFOX 4 Versus FOLFOX 4 Plus Cetuximab Versus Immediate Surgery for High-Risk Stage II and III Colon Cancers: A Phase II Multicenter Randomized Controlled Trial (PRODIGE 22). Ann Surg. 2020 Apr;271(4):637-645. doi: 10.1097/SLA.0000000000003454. PMID 31356278
- [Derived] Karoui M, Rullier A, Luciani A, Bonnetain F, Auriault ML, Sarran A, Monges G, Trillaud H, Le Malicot K, Leroy K, Sobhani I, Bardier A, Moreau M, Brindel I, Seitz JF, Taieb J. Neoadjuvant FOLFOX 4 versus FOLFOX 4 with Cetuximab versus immediate surgery for high-risk stage II and III colon cancers: a multicentre randomised controlled phase II trial--the PRODIGE 22--ECKINOXE trial. BMC Cancer. 2015 Jul 10;15:511. doi: 10.1186/s12885-015-1507-3. PMID 26156156